CLINICAL TRIAL: NCT00036088
Title: Olanzapine Versus An Active Comparator in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2347; F1D-MC-HGHJ
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
The purpose of this study is to determine how Olanzapine compares to an active comparator in the treatment of schizophrenia

ELIGIBILITY:
Inclusion:

1. You must be between the ages of 18 and 75. If you have reached your 76th birthday, you will not be able to participate
2. You must have been diagnosed with schizophrenia
3. You must be able to visit the doctor's office as scheduled for the next 7 months

Exclusion:

1. You have a serious medical illness, such as heart, liver, or kidney disease (Note: If you are uncertain about a particular condition, discuss it with your doctor.)
2. You are either pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 530
Dates: Start 2001-08; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Locations (60):
- United States (25):
  - El Centro, California
  - Glendale, California
  - Sherman Oaks, California
  - Middleton, Connecticut
  - Norwich, Connecticut
  - Melbourne, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Lafayette, Indiana
  - Rockville, Maryland
  - Newton, Massachusetts
  - Saint Charles, Missouri
  - New York, New York
  - Olean, New York
  - Staten Island, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - El Paso, Texas
  - Houston, Texas
  - Terrell, Texas
  - Richmond, Virginia
- Argentina (4):
  - La Plata, Buenos Aires
  - Godoy Cruz, Mendoza Province
  - Buenos Aires
  - Ciudad de Buenos Air
- Austria (5):
  - Graz
  - Innsbruck
  - Linz
  - Wein
  - Wels
- Brazil (5):
  - Salvador, Estado de Bahia
  - Aparecida de Goiânia, Goiás
  - Pelotas, Rio Grande do Sul
  - Sau Paulo, Sau Paulo
  - Rio de Janeiro
- Germany (3):
  - Essen
  - Hamburg
  - Tübingen
- Dublin, Ireland
- Mexico City, Mexico
- Lima, Peru
- Puerto Rico (4):
  - Cidra
  - Ponce
  - Rio Piedras
  - San Juan
- Spain (5):
  - Barcelona, Barcelona
  - San Boi de Llobregat, Barcelona
  - Elizondo, Navarre
  - Pamplona, Navarre
  - Langreo, Principality of Asturias
- United Kingdom (5):
  - Camberwell, London
  - London, London
  - Kings Lynn, Norfolk
  - Paisley, Scotland
  - Guildford, Surrey
- Caracas, Venezuela

REFERENCES:
- [Derived] Liu-Seifert H, Ascher-Svanum H, Osuntokun O, Jen KY, Gomez JC. Change in level of productivity in the treatment of schizophrenia with olanzapine or other antipsychotics. BMC Psychiatry. 2011 May 17;11:87. doi: 10.1186/1471-244X-11-87. PMID 21586165